CLINICAL TRIAL: NCT06877715
Title: Autistic Symptomatology and Sensory Profile in Children With Prader-Willi Syndrome
Acronym: CASSPER
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/24/0447; ID-RCB : 2025-A00085-44 (Other: ANSM)
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Prader-Willi Syndrome
Keywords: Prader-Willi syndrome; Autism Spectrum Disorder; Autistic Symptomatology; Sensory profile
MeSH Terms: conditions — Prader-Willi Syndrome; Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children Aged 3 to 16 Years
  Interventions: Other: psychological and sensorial tests

INTERVENTIONS:
Other: psychological and sensorial tests — children receive questionnaires and sensorial test

SUMMARY:
Prader-Willi Syndrome (PWS) is a rare neurodevelopmental disorder stemming from genetic damage in the 15q11-q13 region, leading to hypothalamic dysfunction. Individuals with PWS often exhibit social interaction challenges, intellectual deficits, significant eating disorders, mood disturbances, and sensory-related autistic features. Although PWS is recognized by DSM-5 as a genetic cause of Autism Spectrum Disorder (ASD), ASD diagnosis in PWS remains rare in France. The CASSPER study aims to investigate the distinct autistic and sensory profiles in children with PWS, also analyzing the potential impact of early oxytocin treatment on these manifestations, in line with recommendations for early and tailored intervention.

DETAILED DESCRIPTION:
Prader-Willi syndrome (PWS) is a rare and complex neurodevelopmental disorder (NDD) with genetic origin linked to chromosomal damage in the 15q11-q13 region and characterised by hypothalamic dysfunction. At the psychiatric level, patients with PWS display difficulties in social interaction, mild to moderate intellectual deficit, major eating disorders, mood disorders and autistic manifestations, including hypo-/hyper-reactivity to sensory stimuli.

While the International Classification (DSM-5) lists PWS as one of the genetic causes of Autism Spectrum Disorder (ASD), little is known about the interaction between autistic traits, sensory features and PWS.

To date, assessment and diagnosis of ASD in PWS remains exceptional in standard care in France, despite the obvious importance of correct assessment for early identification and intervention.

In this context, the CASSPER study aims to identify the specificity of PWS in terms of autistic symptomatology and sensory characteristics. The CASSPER study is in line with the recommendations of the French National Health Authority (HAS) for early and appropriate guidance of children with PWS.

In addition, almost all children with PWS under the age of 5 have received early treatment with oxytocin (OT). As the neuromodulatory effect of OT treatment and the involvement of this neurohormone in the development of attachment, social interaction and sensory processing may explain a difference in autistic symptomatology, this parameter will be included in the analyses.

The CASSPER study aims to fill gaps in our knowledge of PWS and its care and could be useful more generally to improve our understanding of autistic manifestations in NDD of genetic origin.

ELIGIBILITY:
Inclusion Criteria:

* Child with genetically confirmed PWS and identification of genetic subtype;
* Child aged between 3 and 16 years;
* Hospitalisation or multidisciplinary consultation planned for the child's routine follow-up at one of the investigating centres;
* No parental/legal guardian objection.

Exclusion Criteria:

* Change in psychotropic treatment (start, change in dose or discontinuation) in the past 3 months;
* Inability to provide clear information to parents/legal guardian;
* Not covered by social security.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consists of children aged 3 to 16 years who have been diagnosed with Prader-Willi syndrome through genetic confirmation, recruited from several hospital centers in France.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Composite criteria : Autistic Symptomatology in Children with Prader-Willi Syndrome: Prevalence, Symptom Specificity, and Variability by Age and Genetic Subtype | day 1 to day 3
  The tests used are the ADOS-2 and ADI-R tests. The ADOS-2 test is used for evaluating the ASD symptoms. It consists of structured and semi-structured activities designed to assess communication, social interaction, play, and restricted or repetitive behaviors. The best possible score is 0, while the worst possible score is 10.
  The other test is ADI-R. The ADI-R is a structured interview used to assess behaviors and developmental history related to ASD. The responses are scored to evaluate the presence and severity of ASD symptoms, helping to support the diagnosis.

SECONDARY OUTCOMES:
Composite criteria : Characterization of the sensory profile of children with PWS | day 1 to day 3
  The PIPS is a program designed to assess and support sensory processing differences in individuals, particularly those with autism. It helps identify sensory sensitivities and adapt interventions accordingly. The highest score is 140, and each modality has a maximum score of 20.
  The ESA-EA is a sensory assessment tool specifically for individuals with autism.
  The U-Sniff measures olfactory function by testing an individual's ability to identify specific odors.
Composite criteria : Correlation Between Autistic Symptoms, Sensory Profile, and Cognitive-Behavioral Disorders, Including Eating Disorders | day 1 to day 3
  This study examines the correlation between autism disorder/sensory profile assessments (ADOS-2, ADI-R, PIPS, ESA-EA, U-Sniff test) and behavioral/cognitive assessments (Vineland-II, CBCL, Dykens questionnaire, IQ). The Vineland-II is a semi-structured interview assessing autonomy and adaptive skills.
  The CBCL evaluates behavioral problems and social skills using a Likert scale, with T-scores indicating severity across clinical subscales.
  The hyperphagia tool for Prader-Willi Syndrome uses a 5-point Likert scale to rate behaviors, calculating total scores and subscores for Hyperphagic Behavior, Drive, and Severity, along with a specific HQ-CT score for clinical trials. Higher scores indicate more severe symptoms in each tool.
Composite criteria : Assessing the Impact of Autistic Symptomatology and Sensory Profile on Family Burden and Quality of Life | day 1 to day 3
  ZBI measures parents' perception of the burden associated with their child's disability, using a 5-point Likert scale ("0" = never, "4" = almost always). A total score is calculated by summing the 22 items, with higher scores indicating a greater burden.
  IOFS explores the impact of a child's disability on the family's quality of life. Parents rate statements on a 4-point Likert scale ("strongly agree" = 1, "strongly disagree" = 4), and a total score is calculated after reversing scores. Higher scores reflect a greater impact on family quality of life.
Composite criteria : comparison of Autistic Symptomatology, Sensory Profile, and Developmental Profile in 5-7 Year-Old Children: Early OT Treatment vs. Untreated | day 1 to day 3
  "In the 5-7 year age group, comparison of scores and subscores between the early OT-treated children group and the untreated children group regarding:
  The specificity of autistic symptomatology (ADOS-2, ADI-R) Sensory profile (PIPS, ESA-EA, U-sniff test) Behavioral and cognitive profile (Vineland-II, CBCL, Dykens questionnaire, IQ) The impact of the condition (ZBI, IOFS)

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Cabal, Principal Investigator — University Hospital of Toulouse
Locations (1):
- Children Hospital, Toulouse, France